CLINICAL TRIAL: NCT03975374
Title: Efficacy and Safety of Tobradex Eye Drop Suspension vs Tobramycin/Dexamethasone Ophthalmic Suspension
Brief Title: To Study Efficacy and Safety of Tobradex Eye Drop Suspension vs Tobramycin/Dexamethasone Ophthalmic Suspension
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sutphin Drugs (Industry)
Responsible Party: Principal Investigator, Dr. Ajai Prakash, President, Sutphin Drugs
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sutphin T
Record Dates: First submitted 2019-05-29; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Blepharo Conjunctivitis
MeSH Terms: interventions — Tobramycin; Tobramycin, Dexamethasone Drug Combination

STUDY DESIGN:
Intervention Model Description: In group one, patients will be instructed to instill 2 gtt of Tobradex ophthalmic solution for 10 days.
  In group two, patients will be instructed to instill 2 gtt of Tobramycin/dexamethasone solution for 10 days .
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tobramycin/Dexamethasone opthamic Solution (Experimental): This group of randomized patients will be instructed to instill 2 gtt of Tobramycin/Dexamethasone opthamic solution every 6 hours for 10 days
  Interventions: Drug: Tobramycin/dexamethasone opthalmic solution
- Tobradex Opthalmic Solution (Active Comparator): This group of randomized patients will be instructed to instill 2 gtt of Tobradex Opthalmic Solution every 6 hours for 10 days
  Interventions: Drug: Tobradex Opthalmic Solution

INTERVENTIONS:
Drug: Tobramycin/dexamethasone opthalmic solution — To compare efficacy and safety in randomized patients recieving Tobradex versus Tobramycin/Dexamethasone opthamic Solution
  Other Names: Tobradex
  Arms: Tobramycin/Dexamethasone opthamic Solution
Drug: Tobradex Opthalmic Solution — Tobradex Opthalmic Solution
  Arms: Tobradex Opthalmic Solution

SUMMARY:
The objective of the study is to compare and describe efficacy and safety of Tobradex ophthalmic suspension versus generic Tobramycin/dexamethasone Suspension in treatment of Blepharoconjuctivitis through clinical parameters

DETAILED DESCRIPTION:
Evaluation of signs and symptoms during treatment, with a record of individual scores for each parameter; Observation and statistical comparison of drug safety, by recording qualitative and quantitative parameters related to adverse effects occurring during treatment.

ELIGIBILITY:
Inclusion Criteria:

* All potential subjects with symptomatic blepharitis examined to have blepharitis with healthy mental status, able to give consent, with/without co-existing medical conditions will be considered

Exclusion Criteria:

* All subjects with history and/or probable history of allergic reaction to tobramycin/dexamethasone and all subjects who have mental disability and are unable to give direct consent will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Estimated)
Dates: Start 2019-06-15 (Estimated); Primary Completion 2019-07-01 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
Sign and symptoms composite score | 10 days
  The change from baseline in the signs and symptoms score. Global sign and symptom score defined as the total score of lid margin redness (0-3), lid swelling (0-4), bulbar conjunctival redness (0-3), palpebral conjunctival redness (0-3), ocular discharge (0-3), itchy eyelids (0-4), and gritty eyes (0-4).
  The change from baseline to Day 10 (Visit 3 at day 1, day 7 and day 10) in the ocular signs and symptoms composite score. Ocular signs and symptoms were collected for study eyes at each study visit using a 0-4 grading scale, assessed as 0 = none, 1 = minimal/trace, 2 = mild, 3 = moderate, and 4 = severe. The signs and symptoms composite score was the sum of each individual sign or symptom score.

CONTACTS AND LOCATIONS:
Overall Officials: Ajai Prakash, Principal Investigator — Sutphin Drugs
Locations (1):
- Sutphin Drugs, Jamaica, New York, United States

IPD SHARING:
Plan to Share IPD: No